CLINICAL TRIAL: NCT04770662
Title: Obsessive-compulsive Symptoms in Children and Adolescents With Anorexia Nervosa and Possible Correlation With BMI
Brief Title: Obsessive-compulsive Symptoms in Children and Adolescents With Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Lisa Cornelis, Principal Investigator, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDIE01PAIKA2020
Record Dates: First submitted 2021-02-13; First posted 2021-02-25 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Anorexia Nervosa
Keywords: obsessive compulsive symptoms
MeSH Terms: conditions — Anorexia Nervosa | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: A national, academic, interventional study. The data will be acquired through questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- research group (Other): patients who are willing to participate in the study
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Administered Questionnaires:
  * Dutch version of Children's Yale-Brown Obsessive Compulsive Scale (CYBOCS, Goodman W.K. e.a.)
  * Dutch version of Eating Disorder Inventory-3 (EDI-3, David M. Garner)
  * General Questionnaire: demografic , scholar and social information and child psychiatric history
  * Dutch version of the Child Behavior Checklist (CBCL, T.M. Achenbach)
  * Anorectic Behavior Observation Scale (ABOS, Vandereycken W., Universitair Centrum Kortenberg, 1992)

SUMMARY:
The purpose of this study is to determine obsessive-compulsive symptoms and BMI changes in children and adolescents with anorexia nervosa and find out whether there is a group-level correlation between the two. We also investigate a possible link between obsessive compulsive symptoms and the psychological features of eating disorders.

It is a national, academic, interventional study. The data will be acquired through questionnaires.

DETAILED DESCRIPTION:
Children and adolescents with anorexia nervosa show a high psychiatric co-morbidity. In clinical practice, compulsions and compulsive thoughts are frequently reported in children and adolescents with anorexia nervosa. Obsessive compulsive disorder occurs in 19% of patients with anorexia nervosa and anorexia nervosa is seen in 3-17% of female patients with obsessive compulsive disorder.

A precise explanation for this coexistence is still unknown.An underlying genetic correlation and common neuropsychological factors and personality traits are described in the literature as possible explanations. Little is know about the relation between obsessive compulsive symptoms and the psychological features of eating disorders.

It is also unclear whether obsessive compulsive symptoms can be seen as a result of the underweight and weight loss associated with anorexia nervosa and whether these symptoms clear up with weight recovery. Research on this is very limited and shows different results. The aim of this study is to examine obsessive compulsive symptoms and weight change in children and adolescents with anorexia nervosa and to determine whether there is a group-level correlation between the two.

It is a national, academic, interventional study. The data will be acquired through the following questionnaires:

* Questionnaires to be completed by the minor:

  * Dutch version of the Children's Yale-Brown Obsessive Compulsive Scale (CYBOCS, Goodman W.K. e.a., vertaald en bewerkt door Lidewij Wolters en Else de Haan, DAT de Bascule, juni 2012, existing of two parts CY-BOCS Symptom Checklist en CY-BOCS Severity Ratings)
  * Dutch version of the Eating Disorder Inventory-3 (EDI-3, David M. Garner, Nederlandse vertaling door Tatjana van Strien, Hogrefe Uitgevers B.V. Amsterdam, 2014)
* Questionnaires to be completed by the parent or guardian:

  * General questionnaire: personal data, family and school and social information, child psychiatric history
  * Dutch version of the problem part of the Child Behavior Checklist (CBCL, T.M. Achenbach, Nederlandse vertaling door F.C. Verhulst en J. van der Ende, Erasmus MC - Sophia Kinderziekenhuis Rotterdam, 2001)
  * Anorectic Behavior Observation Scale (ABOS, Vandereycken W., Universitair Centrum Kortenberg, 1992)
  * Consent Form to contact if the completed questionnaires have increased results

ELIGIBILITY:
Inclusion Criteria:

* Dutch-speaking female patients with parents who have sufficient command of Dutch
* Minors from 10 years up to and including 18 years old
* Known with the diagnosis of anorexia nervosa and registered for treatment in Paika Food Clinic Service (outpatients and/or inpatients)
* Informed consent obtained from the minor herself and parent (s) / guardian

Exclusion Criteria:

* Patients or parents of patients who do not have sufficient command of Dutch

  * Male patients
  * Minors <10 years and adults older than 18 years
  * Minors and / or parent (s) / guardians have not given written permission to participate

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of obsessive compulsive symptoms | through study completion, an average of 1 year
  current obsessive compulsive symptoms are identified using the CY-BOCS Symptom Checklist (17 different categories of obsessive compulsive behaviour en thoughts, each scored by 0 (if absent) or 1 (if present). A total score is calculated by taking the mean of all 17 categories (=' total number of obsessive compulsive symptoms').
Severity of obsessive compulsive symptoms | through study completion, an average of 1 year
  severity of symptoms are identified using the CY-BOCS Severity Ratings score between minimum value 0 (no impact on daily life) and maximum value 40 (high impact on daily life)

SECONDARY OUTCOMES:
Correlation between the severity and total number of obsessive compulsive symptoms and BMI | through study completion, an average of 1 year
  Correlation between the severity and the total number of obsessive compulsive symptoms using CY-BOCS Severity Ratings, score between minimum value 0 (no impact) and maximum value 40 (high impact) and BMI (in kg/m^2). For BMI we measure 'current BMI' = BMI on the moment of inclusion to the study, 'past BMI' = BMI 6 months before that en 'BMI-change' = the difference between 'past BMI' and 'current BMI'
Correlation between obsessive compulsive symptoms (severity and total number) and EDI-3 subscales | through study completion, an average of 1 year
  Correlation between the severity and the total number of obsessive compulsive symptoms using CY-BOCS Severity Ratings, score between minimum value 0 (no impact) and maximum value 40 (high impact) and EDI-3 subscales. For BMI we measure 'current BMI' = BMI on the moment of inclusion to the study, 'past BMI' = BMI 6 months before that en 'BMI-change' = the difference between 'past BMI' and 'current BMI'. The EDI-3 subscales includes the eating disorder symptoms, i.e., drive for thinness (DT), bulimia (B) and body dissatisfaction (BD) and more general psychological features related to eating disorders i.e. low self-esteem (LSE), personal alienation (PA), interpersonal insecurity (II), interpersonal alienation (IA), interoceptive deficits (ID), emotional dysregulation (ED), perfectionism (P), asceticism (AS) and maturity fear (MF).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No